CLINICAL TRIAL: NCT06772103
Title: Biceps Tenodesis with 360 Suture Anchor Versus Self Locking Tenodesis in the Absence of Rotator Cuff Tears
Acronym: Blast2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Générale dAnnecy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-43-CGA
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: SLAP Lesion
Keywords: biceps; tenodesis; imaging; tendon repair

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- self-locking biceps tenodesis (Experimental)
  Interventions: Procedure: self-locking biceps tenodesis
- 360° double-loop lasso biceps tenodesis (Active Comparator)
  Interventions: Procedure: Biceps Tenodesis with 360 Suture anchor

INTERVENTIONS:
Procedure: self-locking biceps tenodesis — The LHB tendon is detached from its origin at the level of the superior labrum. This technique supports the self-locking mechanism of the LHB tendon in the bicipital groove by detaching the tendon from the Y-shaped superior glenoid, including the superior labrum. A radiographically visible suture will be attached to the proximal part of the LHB tendon to facilitate subsequent localization of the LHB tendon during imaging (3-0 stainless steel, ethicon).
  Arms: self-locking biceps tenodesis
Procedure: Biceps Tenodesis with 360 Suture anchor — The LHB tendon is detached from its origin and sutured. Next, the LHB tendon is fixed in the bicipital groove using a 360-loop tenodesis technique with the Knotless FiberTak® biceps implant system. A radiographically visible suture will be attached to the proximal part of the LHB tendon to facilitate subsequent localization of the LHB tendon during imaging (3-0 stainless steel, ethicon).
  Arms: 360° double-loop lasso biceps tenodesis

SUMMARY:
This is a prospective randomized controlled trial. The aim of this study is to compare the clinical results and complications of self-locking biceps tenodesis and double-loop 360 lasso biceps tenodesis for the treatment of pathology of the long head of the biceps or superior labrum anterior-posterior (SLAP) during shoulder arthroscopy in patients without arthroscopic rotator cuff tears. Currently, there is no consensus on the use of tenodesis versus tenotomy to treat pathology of the long head of the biceps during arthroscopic rotator cuff repair. Numerous studies have examined the clinical results of long biceps tenotomy versus long biceps tenodesis, and there is no evidence to date of superiority of either technique. However, these studies were carried out on patients with rotator cuff tears, and so it has not been possible to directly compare the two procedures. At Clinique Générale, we use a new, innovative technique called autobloc tenodesis to treat pathologies of the long head of the biceps. There are no comparative studies between autobloc tenodesis of the biceps and biceps tenodesis in patients without rotator cuff tears. Given its potential advantages, autobloc biceps tenodesis could become the new technique of choice for treating biceps longus tendon pathology, potentially reducing differences in outcomes such as Popeye deformity. The information provided by this study could potentially guide future clinical practice, helping surgeons choose the most appropriate treatment for their patients with long biceps tendon pathology.

ELIGIBILITY:
Inclusion Criteria:

* Tendinopathy of the Long Head of the Biceps based on clinical symptoms or SLAP-type lesion
* Partial thickness rupture or absence of rupture of the rotator cuff of the subscapular, supraspinatus and/or infraspinatus tendons, diagnosed preoperatively on ultrasound, arthro-CT or MRI.

Exclusion Criteria:

* Osteoarthritis of the glenohumeral joint, defined by narrowing of the glenohumeral joint space or osteophytes, using AP radiography of the affected shoulder.
* Distance between acromion and humeral head measuring 6 mm or less
* Previous shoulder surgery.
* Dementia or inability to complete questionnaires and assessments.
* Pregnant or breast-feeding patient
* Protected adult patient
* Patient not covered by social security.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Constant score | 1 year after surgery
  100-point scale comprising four components, including a patient-reported section (pain 15 points and activity level 20 points), for a total of 35 points. Alongside this is a doctor-reported section (shoulder strength 25 points, range of motion 40 points) for a total of 65 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Générale, Annecy, France

IPD SHARING:
Plan to Share IPD: No